CLINICAL TRIAL: NCT02124447
Title: Comparison of Efficacy and Patient Tolerability of Four Commercially Available Bowel Purgatives for Screening and Surveillance Colonoscopy: A Single Tertiary Medical Center Experience.
Brief Title: Single Center Comparison of 4 FDA Approved, Commercially Available Bowel Purgatives for Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol issues. Modifications potentially will be undertaken and resubmitted to IRB
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Zachary Smith, Division of Gastroenterology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PRO00022505
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Patients Undergoing Screening or Surveillance Colonoscopy
MeSH Terms: interventions — Golytely; MoviPrep; Sulfates

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- PEG+E (Active Comparator): Split dose 4 liter polyethylene glycol with electrolytes
  Interventions: Drug: PEG+E
- PEG+Asc (Active Comparator): Split dose 2 liter polyethylene glycol with ascorbic acid
  Interventions: Drug: PEG+Asc
- P+MC (Active Comparator): Split dose sodium picosulfate, magnesium oxide, and anhydrous citric acid
  Interventions: Drug: P+MC
- sulfate (Active Comparator): Split dose sodium sulfate, magnesium sulfate, and potassium sulfate solution
  Interventions: Drug: sulfate

INTERVENTIONS:
Drug: PEG+E — Split dose 4 liter polyethylene glycol with electrolytes
  Other Names: Golytely
  Arms: PEG+E
Drug: PEG+Asc — Split dose 2 liter polyethylene glycol with ascorbic acid
  Other Names: MoviPrep
  Arms: PEG+Asc
Drug: P+MC — Split dose sodium picosulfate, magnesium oxide, and anhydrous citric acid
  Other Names: Suprep
  Arms: P+MC
Drug: sulfate — Split dose sodium sulfate, magnesium sulfate, and potassium sulfate solution
  Other Names: Prepopik
  Arms: sulfate

SUMMARY:
This will be a 4-way comparison to prospectively evaluate the efficacy and patient tolerability of four commercially available bowel preparations among patients undergoing colonoscopy for screening and surveillance in a single tertiary academic medical center.

DETAILED DESCRIPTION:
We will randomize 300 consecutive patients undergoing colonoscopy for screening or surveillance purposes to receive one of four bowel purgatives. These purgatives include

1. Split dose 4 liter polyethylene glycol with electrolytes (PEG+E): Brand name GoLytely
2. Split dose 2 liter polyethylene glycol with ascorbic acid (PEG+Asc): Brand name: MoviPrep
3. Split dose sodium picosulfate, magnesium oxide, and anhydrous citric acid (P+MC): Brand name Prepopik
4. Split dose sodium sulfate, magnesium sulfate, and potassium sulfate solution (sulfate): Brand name Suprep

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater
2. Ability to understand and complete questionnaires
3. Ability to speak and read English
4. Willingness to participate in study
5. Colonoscopy is being performed for routine screening (i.e. no prior personal history of polyps or cancer) or surveillance (i.e. follow up for a personal history of polyps) purposes

Exclusion Criteria:

1. Previous bowel resection of any kind (small or large bowel)
2. End stage renal disease (ESRD)
3. Contraindication to bowel purgative
4. Necessity for inpatient admission to receive bowel preparation for any reason
5. Currently taking any narcotic/opiate pain or anticholinergic medication (since these may predispose to higher colon stool burden at baseline)
6. Currently taking stool softeners (e.g. Miralax, Amitiza, Linzess, lactulose) or stimulant laxatives (e.g. Dulcolax)
7. Subject did not follow appropriate dosing instructions for bowel purgative
8. Colonoscopy is being performed to evaluate a clinical symptom such as rectal bleeding, constipation, abdominal pain, or diarrhea
9. History of colon polyposis syndrome
10. Personal history of inflammatory bowel disease
11. History of inadequate colon preparation on any prior colonoscopies
12. Patient is pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of bowel cleansing according to the Boston Bowel Preparation Score (BPPS) | Patient outcome will be assessed at the time of the colonoscopy by the performing physician and ducomentation of this outcome will occur within 24 hours of the procedure

SECONDARY OUTCOMES:
Patient tolerability and satisfaction | Outcome of satisfaction will be assessed on a single survey that the patient will provide the day of their colonoscopy and will be recorded by study personnel up to 30 days thereafter
  Will be assessed using a previously studied satisfaction questionnaire (7 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital & The Medical College of Wisconsin, Milwaukee, Wisconsin, United States